CLINICAL TRIAL: NCT02468622
Title: Transcriptomic and Biochemical Changes During Spontaneous Attacks of Migraine With Aura and Migraine Without Aura
Brief Title: Transcriptomic and Biochemical Changes During a Migraine Attack
Status: Completed | Type: Observational
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Katrine Falkenberg, Medical doctor, Danish Headache Center
Other Study IDs: Transcriptomics
Record Dates: First submitted 2015-06-04; First posted 2015-06-11 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2019-12

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bloodsamples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- MO patients: Patients with migraine without aura. We will take blood samples during spontaneous migraine attacks
  Interventions: Other: Blood samples
- MA patients: Patients with migraine with aura. We will take blood samples during spontaneous migraine attacks
  Interventions: Other: Blood samples

INTERVENTIONS:
Other: Blood samples — There is no intervention, but we will take blood samples during a spontaneous migraine attack

SUMMARY:
Despite the fact that migraine is a common disorder, the pathogenesis is still not fully elucidated. Studying transcriptomic and biochemical changes during induced and spontaneous migraine-attacks will enhance our understanding and may point to new targets for drug development.

DETAILED DESCRIPTION:
Migraine is a common neurological disorder affecting approx. 16 % of the European population. Despite the fact that migraine is a common disorder, the pathogenesis is still not sufficiently known.

Studying transcriptomic and biochemical changes during spontaneous migraine-attacks will greatly enhance our understanding of migraine mechanisms and may point to new targets for drug development.

Two blood samples (one for RNA analysis and one for biochemical analysis) are taken on minimum 15 patient with migraine with aura and 15 patients with migraine without aura when they experience a spontaneous migraine attack. A second sample is taken 2 hours after treatment with subcutaneous sumatriptan. Another two blood samples are taken when the patient has been migraine free for at least 5 days and had no other headache for at least 24 hours. A fourth set of blood samples are collected after a cold pressor test.

ELIGIBILITY:
Inclusion Criteria:

* Migraine patients who meet IHS criteria for migraine with or without aura of both sexes,
* 18-70 years,
* 45-95 kg.

Exclusion Criteria:

* any other type of headache then migraine without aura (except episodic tension-type headache < 1 day per week),
* serious somatic or psychiatric disease,
* pregnancy,
* and intake of daily medication (except oral contraceptives).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 15 patients with migraine without aura and 15 paitients with migraine with aura
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2015-08; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Transcriptomic changes | 2 year
  The investigators will measure transcriptomic changes using Next Generation Sequencing during a migraine attack
Changes in CGRP levels during a migraine attack (CGRP1-37, CGRP1-17, CGRP18-37, CGRP1-26, CGRP27-37) | 2 year
  The investigators will use advanced mass spectrometry to measure CGRP levels
Changes in PACAP levels during a migraine attack (PACAP-27, PACAP-38 ) | 2 years
  The investigators will use advanced mass spectrometry to measure PACAP levels
Changes in VIP, glutamate, serotonin, PGE-2, nitric oxide metabolites, cAMP, and cGMP | 2 years
  The investigators will use advanced mass spectrometry to measure VIP, glutamate, serotonin, PGE-2, nitric oxide metabolites, cAMP, and cGMP during a migraine attack
Changes in Metabolomics | 3 years
  The investigators will use advanced mass spectrometry (LC-MS) to measure metabolomics in the 4 blood samples
Changes in Proteomics | 3 years
  The investigators will use advanced mass spectrometry to measure proteomics in the 4 blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Emma Katrine Hansen, Doctor, Principal Investigator — Danish Headache Center
Locations (1):
- Emma Katrine Hansen, Copenhagen, Glostrup, Denmark